CLINICAL TRIAL: NCT03645486
Title: Lentiviral Gene Therapy for Chronic Granulomatous Disease (CGD)
Brief Title: Lentiviral Gene Therapy for CGD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-18004
Record Dates: First submitted 2018-07-24; First posted 2018-08-24 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Chronic Granulomatous Disease
Keywords: Chronic granulomatous disease; Lentiviral vector
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lentiviral TYF-CGD-modified autologous stem cells (Experimental): Autologous hematopoietic stem cells transduced with lentiviral TYF vector carrying the functional gene
  Interventions: Genetic: Infusion of lentiviral TYF-CGD-modified autologous stem cells

INTERVENTIONS:
Genetic: Infusion of lentiviral TYF-CGD-modified autologous stem cells — Infusion of lentiviral TYF-modified autologous stem cells at 1~10x10^6 gene-modified cells per kg body weight

SUMMARY:
This is a Phase I/II clinical trial of gene therapy for treating Chronic Granulomatous Disease using a high-safety, high-efficiency, self-inactivating lentiviral vector TYF to functionally correct the defective gene. The objectives are to evaluate the safety and efficacy of the TYF-CGD gene transfer clinical protocol.

DETAILED DESCRIPTION:
Chronic granulomatous disease (CGD) is a rare disorder caused by inherited defects in the NADPH oxidase multienzyme complex. It is associated with severe and life-threatening bacterial and fungal infections. Approximately two-thirds of all CGD cases result from mutations within the X-linked gp91phox gene (CYBB), followed by the autosomal recessive forms of CGD, with defects in the gene coding for p47phox (NCF1) accounting for 10-30% of all CGD cases.

The primary objectives are to evaluate the safety of the advanced self-inactivating lentiviral vector TYF-CYBB and TYF-NCF1, the ex-vivo gene transfer clinical protocol and the efficacy of immune reconstitution in patients overcoming frequent infections present at the time of treatment, assessment of vector integration sites, and finally the long-term correction of immune dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

1. CGD patients >= 0 years of age
2. Molecular diagnosis confirmed by DNA sequencing and supported by laboratory evidence for absent or significantly reduced biochemical activities of the NADPH-oxidase
3. Karnofsky-Index > =70%
4. At least one prior, ongoing or refractory severe infection and/or inflammatory complications requiring hospitalization despite drug intervention
5. Written informed consent for adult patient, and assent for pediatric subjects seven years or older

Exclusion Criteria:

1. Contraindication for leukapheresis (anaemia Hb <8g/dl, cardiovascular instability, severe coagulopathy) or for administration of conditioning medication
2. Female patients who are pregnant or lactating as determined by history and/or positive pregnancy test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 15 year follow up
  Patient will be monitored for overall health condition, including immune cell assessments, blood biochemistry and metabolitic activities, metabolic detoxification.
Gene marking in bone marrow cells | 15 year follow up
  Gene-modified cells in the bone marrow will be measured by vector-specific quantitative PCR of colony-forming cells. Patient overall survival will be followed up for 15 years.

SECONDARY OUTCOMES:
Change in infection frequency | 1 year after treatment by clinical history, complete physical examination, haematological and microbiological tests
Recovery of immune function | 1 year follow up
  Whole blood cell counts (WBC), including CD3+ CD4, CD8 T cells, CD19+ B cells and CD16/CD56 NK cells, and absolute neutrophil counts (ANC), the percentage of NADPH oxidase positive cells, and the kinetics of transduced cells as determined by dihydrorhodamine (DHR) assay, will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No